CLINICAL TRIAL: NCT06652347
Title: Facilitating the Engagement and Satisfaction of Older Adults in Their Cancer Care Planning: A Randomized Study to Understand the Preferences and Views of Older Adults Regarding the Use of Geriatric and Objective Functional Assessments for Cancer Treatment Planning
Brief Title: Understanding the Preferences and Views of Older Adults on the Use of Geriatric and Objective Functional Assessments for Cancer Treatment Planning.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Zachary Frosch, Assistant Professor Department of Hematology/Oncology, Fox Chase Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-1020
Record Dates: First submitted 2024-10-15; First posted 2024-10-22 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Care Delivery; Geriatrics; Geriatric Assessment
Keywords: fitness tracking; Care delivery Intervention; Functional Status in Older Adults; Cancer Treatment Preferences; Quality vs Quantity of Life; Patient-Reported Outcomes in Oncology; Randomized Controlled Trial; Quality of Life in Cancer care; Functional Health Assessments; Patient-Centered Cancer Treatment
MeSH Terms: interventions — Aging; Surveys and Questionnaires; Body Modification, Non-Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Sharing Arm (Experimental): early sharing of GA and OFS results to participants
  Interventions: Other: Cancer care delivery
- Delayed Sharing Arm (No Intervention): delayed sharing of GA and OFS results to participants

INTERVENTIONS:
Other: Cancer care delivery — Early vs. delayed sharing of GA and OFS diagnostic results and how that sharing affects patient preferences, decision- making, and satisfaction in the context of participants' cancer care.
  Other Names: geriatric and OFS assessment; Quality Quantity (QQ) questionnaire; Non-therapeutic
  Arms: Early Sharing Arm

SUMMARY:
This Interventional clinical study aims to explore how receiving information about their health and physical abilities affects the treatment decisions of older adults. The study will look at whether sharing detailed assessments of their health and functional status helps older adults better understand their condition and make informed decisions about their care.

The main question it aims to answer is if providing this information changes the treatment priorities of older adults, helping them focus on what matters most to them in their medical care.

DETAILED DESCRIPTION:
This randomized, interventional, cancer care delivery trial will test whether receipt of Geriatric Assessment (GA) and Objective Functional Status (OFS) assessment data affects older adults' treatment priorities. It will also assess the preferences of older adults for the collection, sharing, and use of their assessment data. Finally, it will explore whether less fit patients experience a lower level of satisfaction and a greater degree of regret with their decision to undergo anti-cancer therapy. This study will utilize a randomized design where participants will be randomized to either the intervention arm (early sharing of GA and OFS results) or to the control arm (delayed sharing of GA and OFS results). To assess patients' preferences for quality vs quantity of life, the investigators will use the Quality Quantity (QQ) questionnaire. All patients will complete this at baseline and then undergo their GA and OFS assessments. Patients randomized to the intervention group will be provided the results of their GA and OFS assessments, and then complete the QQ Questionnaire for a second time to assess for any changes following receipt of their assessment results. Patients randomized to the control group will undergo the assessments and complete the same questionnaire as the intervention group but will not receive the results of their GA and OFS assessments prior to completing the second QQ Questionnaire. For the control group, assessment results will be shared with patients after completion of the follow-up QQ Questionnaire. After reviewing their assessment results, patients in both groups will then complete a questionnaire that inquire about their preferences for receipt, use, and sharing of their assessment data. It will also inquire about the degree to which receipt of these data affected how they experienced their cancer care.

The Investigators will determine whether sharing of geriatric and OFS assessment results affected patients' treatment priorities by measuring the absolute change from baseline in the QQ questionnaire scores for quantity and quality of life, comparing the change in the intervention versus the control group. The Investigators will also describe patients' preferences for the collection, use and sharing of their assessment data as reported in the preferences questionnaire, both overall and by race/ethnicity. To explore differences in patients' satisfaction with their decision to pursue anti-cancer therapy by functional status level, participants will complete the "Was it Worth It" (WIWI) questionnaire at the first of either 1) the conclusion of their treatment regimen or 2) three months after enrollment. The provider assessment will ask whether patients experienced any of the following: a toxicity of treatment ≥grade 3, treatment dose reduction, treatment interruption, treatment discontinuation, hospitalization, or a decline in performance status.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65

At the time of study screening either:

* Started a new qualifying index regimen within the last 30 days (inclusive)
* Are being considered for a new qualifying index regimen

Exclusion Criteria:

* Patients will be excluded if they

  * Do not have the capacity to consent to study procedures
  * Are unable to complete English language questionnaires
  * Are already using an activity tracker on a daily basis (and therefore may be aware of their current level of activity)
  * Are enrolled in another study in which physical activity is a substantial part or all of the therapeutic intervention or where physical activity is specifically being evaluated and shared with patients. Patients on studies not evaluating or sharing physical activity are eligible for the present study if they meet the other inclusion/exclusion criteria and participation in the present study is not excluded by other studies in which they are enrolled.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Absolute change in QQ-Length of life from baseline to post-intervention | From baseline questionnaire at enrollment to post intervention questionnaire at an average of 4 weeks after enrollment.
  The QQ uses a 5-point Likert scale to rate each of the 4 questions on the QQ-L subscale. The scores for this subscale are then summed, meaning that patients will receive a score ranging from 4-20 for the QQ-L. The total score from the 4 QQ-L items measures the strength of a participant's preference for length of life, with higher scores meaning greater preference for length of life.

SECONDARY OUTCOMES:
The secondary outcome will be the absolute change in the QQ quality of life subscale (QQ-Q) from baseline to post-intervention. | From baseline questionnaire at enrollment to post intervention questionnaire at an average of 4 weeks after enrollment.
  The QQ uses a 5-point Likert scale to rate each of the 4 questions on the QQ-Q subscale. The scores for the subscale are then summed, meaning that patients will receive a score ranging from 4-20 for the QQ-Q. The total score from the 4 QQ-Q items measures the strength of a participant's preference for quality of life, with higher scores meaning greater preference for quality of life.

OTHER OUTCOMES:
The proportion of patients who, on the Was It Worth It (WIWI) questionnaire, report that their treatment was worthwhile, that they would undergo it again, and that they would recommend it to others. | From enrollment to the end of treatment or at 3 months after study entry, whichever comes first.
  The proportion of patients who, on the Was It Worth It (WIWI) questionnaire, report that their treatment was worthwhile, that they would undergo it again, and that they would recommend it to others.
Summary/descriptive statistics for participants' answers to the preferences questionnaire. | From baseline questionnaire at enrollment to post intervention questionnaire at an average of 4 weeks after enrollment.
  It inquires about their preferences for receipt, use and sharing of their assessment results, along with the degree to which receipt of these results affected their understanding or approach to their care

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Frosch, MD, MSHP, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared due to privacy concerns.